CLINICAL TRIAL: NCT05877560
Title: A Randomized Controlled Study Using Non-invasive Brain Stimulation to Facilitate the Effectiveness of Vergence/Accommodative Therapy in Symptomatic Convergence Insufficiency
Brief Title: Non-invasive Brain Stimulation for Treating Symptomatic Convergence Insufficiency
Acronym: NIBSCI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Midwestern University (Other)
Responsible Party: Principal Investigator, Arijit Chakraborty, Assistant Director of Research, Midwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CIRB-IL 22013
Record Dates: First submitted 2023-05-17; First posted 2023-05-26 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Convergence Insufficiency
Keywords: Convergence Insufficiency; Non-invasive Brain Stimulation; Office-Based Vergence/Accommodative Therapy; Frontal Eye Fields; Transcranial Direct Current Stimulation
MeSH Terms: conditions — Ocular Motility Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- NIBS-OBVAT (Active Comparator): 8 sessions of non-invasive brain stimulation with 8 weeks of office-based vergence/accommodative therapy.
  Interventions: Device: Anodal-Transcranial Direct Current Stimulation; Behavioral: Office-Based Vergence/Accommodative Therapy
- NIBS (Active Comparator): 8 sessions of non-invasive brain stimulation only.
  Interventions: Device: Anodal-Transcranial Direct Current Stimulation
- OBVAT (Sham Comparator): 8 sessions of sham stimulation with 8 weeks of office-based vergence/accommodative therapy.
  Interventions: Behavioral: Office-Based Vergence/Accommodative Therapy; Device: Sham Transcranial Direct Current Stimulation

INTERVENTIONS:
Device: Anodal-Transcranial Direct Current Stimulation — Non-invasive brain stimulation will involve the use of anodal transcranial direct current stimulation to apply a 2 milliamp current over the left frontal eye field for approximately 20 minutes with a ramp up to the maximum programmed current and ramp down of 20 seconds.
  Other Names: tDCS; a-tDCS
  Arms: NIBS; NIBS-OBVAT
Behavioral: Office-Based Vergence/Accommodative Therapy — Office-based vergence accommodative therapy involves weekly in-office appointments with the therapist lasting approximately 60 minutes per visit during which time in-office procedures will be performed, and home therapy procedures will be demonstrated. Participants will be prescribed 15 minutes of home reinforcement therapy procedures to be completed 5 days per week. Therapy will consist of two phases adapted from the Convergence Insufficiency Treatment Trial (CITT). Therapy procedures will include gross convergence, accommodation. non-computer based vergence, and computer-based vergence.
  Other Names: OBVAT; Orthoptic training
  Arms: NIBS-OBVAT; OBVAT
Device: Sham Transcranial Direct Current Stimulation — Sham transcranial direct current stimulation will be applied over the left frontal eye field with the current ramping up for 20 seconds before ramping down for 20 seconds. The 2 milliamp current stimulation will occur for only a few seconds at the start and at the end of the 20 minutes.
  Other Names: Sham tDCS
  Arms: OBVAT

SUMMARY:
The goal of this randomized controlled trial is to test the effectiveness of non-invasive brain stimulation in treating adults with symptomatic convergence insufficiency compared to vergence/accommodative therapy. The main questions it aims to answer are:

1. Can non-invasive brain stimulation shorten the treatment time of office-based vergence/accommodative therapy for convergence insufficiency?
2. Is non-invasive brain stimulation alone just as effective as office-based vergence/accommodative therapy in treating convergence insufficiency?

The investigators hypothesize that non-invasive brain stimulation will shorten the treatment time from 12 weeks to 8 weeks of office-based vergence/accommodative therapy and that non-invasive brain stimulation alone would be equally effective as office-based vergence/accommodative therapy in improving symptomatic convergence insufficiency.

Participants will be randomized into one of three treatment groups:

1. Non-invasive brain stimulation with office-based vergence/accommodative therapy.
2. Sham stimulation with office-based vergence/accommodative therapy.
3. Non-invasive brain stimulation only.

Researchers will compare baseline measurements of near point of convergence (NPC) and positive fusional vergence (PFV) to post-treatment measurements for each group.

ELIGIBILITY:
Inclusion Criteria:

* Best-corrected visual acuity of > 20/25 in each eye at distance and near
* Exophoria at near at least 4∆ greater than at far
* Receded near point of convergence of > 6 cm break
* Insufficient positive fusional vergence at near (< 15∆ base-out blur or break)
* CISS score of 16 and greater for children or 21 and greater for adults
* Have had a dilated fundus examination within the last 12 months
* Informed consent and willingness to participate in the study and be randomized

Exclusion Criteria:

* Previously treated for convergence insufficiency with home- or office-based vergence/accommodative therapy
* Amblyopia (> 2-line difference in best-corrected visual acuity between the two eyes)
* Constant strabismus
* History of strabismus surgery
* Convergence insufficiency secondary to acquired brain injury or neurological disorder
* Manifest or latent nystagmus
* Systemic disease known to affect accommodation, vergence, and ocular motility including multiple sclerosis, Graves disease, myasthenia gravis, Parkinson's disease, cerebral palsy, and diabetes
* Developmental disability, attention deficit hyperactivity disorder (ADHD), learning disability or cognitive dysfunction that would interfere with treatment
* Taking medications that can affect normal neurological function including antipsychotics, antiepileptics, and opioids
* Presence of metal or electronic implants in or on the body, including pacemakers

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Near Point of Convergence (NPC) | 4 weeks, 6 weeks, and 8 weeks during treatment; 6 months and 12 months post-treatment
  A change in the NPC break and recovery values measured in centimeters (cm) from baseline after treatment.
Positive Fusional Vergence (PFV) | 4 weeks, 6 weeks, and 8 weeks during treatment; 6 months and 12 months post-treatment
  A change in the near PFV blur, break, and recovery values measured in prism diopters (∆) from baseline after treatment.

SECONDARY OUTCOMES:
Convergence Insufficiency Symptoms Survey (CISS) | 8 weeks during treatment; 6 months and 12 months post-treatment
  A change in the CISS score from baseline after treatment. The minimum score is 0 and the maximum score is 60. Lower scores indicate a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Midwestern University Eye Institute, Downers Grove, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Duval JL, Jaubert D, Poizot-Martin I, De Jaureguiberry JP, Lafeuillade A, Giovannini M, Carloz E, Dhiver C, Gastaut JA. [Colonic leishmaniasis in AIDS]. Ann Med Interne (Paris). 1994;145(3):198-9. No abstract available. French. PMID 8092638
- [Background] Xie Y, Wan B, Li W. [Effect of bee pollen on maternal nutrition and fetal growth]. Hua Xi Yi Ke Da Xue Xue Bao. 1994 Dec;25(4):434-7. Chinese. PMID 7744390
- [Background] Nakano H, Ida T, Harada A, Horiba K, Sakakibara T, Kawase M, Tatsuno K, Obunai Y, Murata M. [Application of epicardial approach technique to the anterior-paraseptal type Wolff-Parkinson-White syndrome]. Kyobu Geka. 1989 May;42(5):358-62. Japanese. PMID 2779032